CLINICAL TRIAL: NCT07070336
Title: The Effect Of Neuroathletic Exercise On Walking Speed, Fall Risk And Cognitive Functions In The Elderly
Brief Title: Neuroathletic Exercise In The Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0001
Record Dates: First submitted 2025-05-26; First posted 2025-07-17 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy Aging
Keywords: aging; neuroathletic exercise; walking speed; gait speed; fall risk; cognitive function

STUDY DESIGN:
Intervention Model Description: The study consists of an experimental and control group. After the pre-tests are applied to the individuals in the experimental groups, neuroathletic exercises will be performed 3 days a week for 12 weeks. Exercises will be performed with the help of a physiotherapist at the KTO Karatay University laboratory 2 days a week, and they will be asked to do it as a home program 1 day a week. At the end of 12 weeks, the final test will be applied and evaluated. The preliminary tests of the control panel are organized as the Activity in the Elderly section of the Activity Guide in Türkiye. During this process, confirmation is collected by frequently calling whether they do any activity outside of their daily routine activities. At the end of 12 weeks, the final test will be applied and the results will be supported with the exercise group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroathletic exercise group (Experimental): After warm-up and reset exercises, eye muscle training will begin with a star chart. Then, it consists of exercises that regulate the accommodation reflex, balance the right and left lobes, regulate the vestibular system, and rhythm exercises.
  After explaining the purpose of the study to the individuals who will be given exercises according to the randomization order, the first measurements will be taken and the exercises will begin. At the end of the 12th week, the measurements will be taken again and the effectiveness of the exercises will be evaluated. The exercises will be done with a physiotherapist 2 days a week, and will be given as a home exercise program for 1 day.
  Interventions: Other: Neuroathletic exercise
- Control Group (No Intervention): Within the scope of the research, after the purpose of the study is explained to the individuals in this group, pre-tests will be conducted according to the randomization order. The individuals in this group will be given the 'Physical Activity in the Elderly' section of the Turkish Physical Activity Guide.

INTERVENTIONS:
Other: Neuroathletic exercise — After warm-up and resetting exercises, it will start with eye muscle training with a star chart. It then consists of exercises that regulate the accommodation reflex, balance the right and left lobes, regulate the vestibular system and rhythm exercises.
  Arms: Neuroathletic exercise group

SUMMARY:
Objective: The aim of this protocol study was to investigate the effect of neuroathletic exercise on walking speed, fall risk and cognitive function in the elderly.

Method: The study is planned as a single-centre, double-blind, parallel group randomised controlled experimental design and will be conducted in accordance with SPIRIT. The sample of the study will consist of healthy elderly people aged 60-80 years. In order to ensure parametric conditions, the sample will be divided into two groups as experimental group (n=30) in which neuroathletic exercise will be performed and control group (n=30) in which Turkey Physical Activity Guidelines will be given and a total of 60 elderly people will be randomly assigned to the groups. The elderly assigned to the experimental and control groups according to the order of randomisation will be administered the timed up and go test (TUG), short physical performance battery (SPPB), geriatric depression scale (GDÖ), MoCA test as pre-test and post-test. The experimental group will be asked to perform neuroathletic exercises two days a week for 12 weeks under the supervision of a physiotherapist, and will be asked to perform a home exercise programme one day a week. The control group will be given the Turkish Physical Activity guide. Data will be collected by the researcher.

Results: Considering the limited number of studies on the use of neuroathletic exercises in the literature, it is thought that our randomised controlled study designed to determine the effect of neuroathletic exercise on walking speed, fall risk and cognitive functions in the elderly will contribute to the literature.

DETAILED DESCRIPTION:
Neuroathletic exercise is an umbrella term encompassing the disciplines of athletic training and neuroscience. The term refers to the further development of biomechanically controlled and defined athletic training through components of movement control by the nervous system. In the early 2000s, athletic trainer Eric Cobb began to combine the two disciplines of athletic training and neuroscience and began to develop a neuroathletic exercise training system for trainers and therapists based on neuroscientific findings. Finally, Cobb combined findings from neuroscience with practical experience from therapy and training to create his own training concept, the Z-Health Performance Training System. The aim of the Z-Health Performance Training System was to integrate movement control systems into classical athletic training, which until then had been completely biomechanically controlled and designed. Neuroathletic training works like this: for every movement perform, the brain needs sensory information from the three movement control systems: the eyes (visual system), balance (vestibular system) and self-perception in space (proprioceptive system). The three movement control systems are very important for neuroathletic exercise. The three movement control systems are very important for neuroathletic exercise. The clearer and better the quality of the signals from these systems, the better the physical performance, and if the communication between the systems is disrupted or the information is too poor, this will negatively affect the success of the exercise. Exercise that focuses on these processes and the weak points of the nervous system is called neuroathletic exercise. It helps to streamline these processes to improve performance and prevent injury. Neuroathletic exercise can help the body regain its ability to process original stimuli and thus improve our quality of life and performance in almost all areas of sport and daily life.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 60-80
* Volunteering to participate in the study
* Having the ability to perform physical, cognitive and sensory tests and exercises

Exclusion Criteria:

* Having a history of injury to the lower and upper extremities within the last year
* Having regular physical activity or sports habits.
* Having participated in any physical activity program in the last 6 months
* Having a sensory pathology that prevents participation in the study
* Having any musculoskeletal, neurological, respiratory or cardiovascular pathology that will limit exercise
* Having a history of malignant disease
* Having an eye defect that cannot be corrected with lenses, such as cataracts, that prevents tests

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Walking speed | 12 week
  • 4-Meter Walking Speed Test: Allows the calculation of walking speed according to the time the participant walks 4 meters on a flat surface. It is a reliable scale widely used to predict mobility and fall risk in elderly individuals (Mehmet et al., 2020)
Fall risk | 12 week
  • Time Up and Go (TUG) Test: It evaluates the functional mobility level and fall risk by measuring the time it takes for the participant to get up from the chair and walk 3 meters, turn around, come back and sit down again in seconds (Podsiadlo et al., 1991).
Cognitive function | 12 week
  • Montreal Cognitive Assessment Scale (MoCA): It is a valid and reliable scale that evaluates the participants' performance in cognitive areas such as executive functions, attention, memory, language, and visual-spatial skills. The total score is evaluated out of 30, and scores of 26 and above are considered normal cognitive levels (Nasreddine et al., 1991).

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is planned to write a report and article with the data of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 year

REFERENCES:
- [Background] Evers J, Stolz I, Klein M. Neuroathletic training in stroke rehabilitation? A single-blind randomized controlled pilot study on the potential of neuroathletic training for balance ability in stroke outpatient rehabilitation. BMC Res Notes. 2024 Dec 12;17(1):358. doi: 10.1186/s13104-024-07022-0. PMID 39668364
- [Background] Lienhard, L., Schmid-Fetzer, U., & Cobb, E. (2019). Neuronale Heilung: Mit einfachen Übungen den Vagusnerv aktivieren-gegen Stress, Depressionen, Ängste, Schmerzen und Verdauungsprobleme. Riva Verlag.
- [Background] Broglio SP, Register-Mihalik JK, Guskiewicz KM, Leddy JJ, Merriman A, Valovich McLeod TC. National Athletic Trainers' Association Bridge Statement: Management of Sport-Related Concussion. J Athl Train. 2024 Mar 1;59(3):225-242. doi: 10.4085/1062-6050-0046.22. PMID 38530653
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10976337/